CLINICAL TRIAL: NCT07319208
Title: Efficacy of Early Continuous Infusion of Hypertonic Saline Solution on the Neurological Outcome at 6 Months in Traumatic Brain Injured Patients. A Single-blinded, Multicenter, Randomized, Controlled Clinical Trial With Blinded Evaluation of the Primary Outcome.
Brief Title: Efficacy of Early Continuous Infusion of HSS on the Neurological Outcome at 6 Months in TBI Patients.
Acronym: COSMOS-TBI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC24_0543; 2024-520205-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-01; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: TBI Traumatic Brain Injury
Keywords: Traumatic brain injury; Saline Solution; Hypertonic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Controlled, Single insulated with blinded assessment of the primary endpoint, Prospective
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Saline Solution (Experimental): Continuous infusion of HSS (NaCl 20%) for 48 hours (can be prolonged during the period of intracranial hypertension)
  Interventions: Drug: Hypertonic saline solution
- Standard (No Intervention): Standard of care

INTERVENTIONS:
Drug: Hypertonic saline solution — Continuous infusion of HSS (NaCl 20%) for 48 hours (can be prolonged during the period of intracranial hypertension)
  Arms: Hypertonic Saline Solution

SUMMARY:
The purpose of this study is to demonstrate the efficacy of early continuous intravenous infusion of hypertonic saline solution (HSS) to improve survival and independence in daily life activities (at 6 months) of patients with traumatic brain injury at high risk of intracranial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to intensive care unit
* Traumatic brain injury with Glasgow Coma Scale ≤ 12
* Intracranial pressure (ICP) monitoring based on the attending physician's clinical judgment, in accordance with guidelines or clinical/radiological signs considered at risk of intracranial hypertension
* Inclusion during the first 12 hours after Intracranial pressure monitoring placement
* Informed and signed consent
* National health insurance

Exclusion Criteria:

* Glasgow Coma Scale (score = 3) and persistent abnormal pupillaryreactivity despite urgent therapy
* Associated cervical spinal cord injury
* Imminent death and do-not-resuscitate orders
* Coma secondary to cardiac arrest
* Pregnancy (serum or urine test performed in routine care)
* Severe Cardiac insufficiency
* Severe chronic renal insufficiency
* Severe hepatic insufficiency: patient presenting with oedemato-ascitic decompensation of liver cirrhosis or patient with Child-Pugh class C cirrhosis
* High risk of follow-up difficulties after ICU discharge
* Patients under court protection
* Patient who does not speak French

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of early continuous of HSS | 3 months
  Survival : number of patients still alive
Efficacy of early continuous of HSS | 6 months
  Rate of moderate to no dependency in activities in daily living at 6 months is defined as a Barthel Index of independence in activities in daily living ≥ 61.

SECONDARY OUTCOMES:
Treatment of intracranial hypertension | 7 days
  Evolution of blood sodium level
Treatment of intracranial hypertension | 7 days
  Evolution of blood chloride level
Treatment of intracranial hypertension | 7 days
  Evolution of solute concentration in blood plasma
Neurological recovery | 7 days
  Number of therapeutic interventions with the TIL (Therapeutic Intensity Level) scale.
Neurological recovery | until 12 months
  Survival : number of patients still alive
Quality of life | until 12 month
  Score of EQ-5D-5L (5-level EuroQol-5D version) : minimum - maximal values: 1-5, higher scores mean a worse outcome.
Quality of life | until 12 months
  Rates of patient living at home, at rehabilitation centers or at hospital
Anterograde amnesia | until 6 months
  Galveston Orientation and Amnesia Test (G.O.A.T) : minimum - maximal values: 0-100, higher scores mean a better outcome.
Neurocognitive functioning | 6 months
  Montreal Cognitive Assessment (MOCA) : minimum - maximal values: 0-30, higher scores mean a better outcome.
Neurological outcome | 6 months
  Glasgow Outcome Scale Extended (GOS-E) : minimum - maximal values: 1-8, higher scores mean a better outcome.
Tolerance | 1 month
  Rates severe hypernatremia (Na> 160 mmol/L)
Tolerance | 1 month
  Rates of acute kidney injury
Tolerance | 1 month
  Number of thrombotic events
Tolerance | 1 month
  Number of entral-pontine myelinolysis
Cost-effectiveness analysis | 12 months
  Incremental cost-effectiveness ratio
Genetic biomarkers | 12 months
  Single nucleotide polymorphism

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHU Caen Normandie, Caen
  - CHU de Clermont- Ferrand, Clermont-Ferrand
  - Hôpital BEAUJON APHP, Clichy
  - CHU Henri Mondor APHP, Créteil
  - CH de Annecy Genevois, Épagny
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - HCL, Lyon
  - AP-HM, Marseille
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU Lariboisière, AP-HP, Paris
  - GHU Paris Cité, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de St- Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided